## STATISTICAL ANALYSIS

The data to be collected for the study will be recorded using SPSS 22 program and analyzed in the same program. Frequency, percentage, mean value, standard deviation, maximum and minimum (min-max) values will be used for descriptive statistics, Pearson Chi square test will be applied for statistical analysis of categorical data and Fisher's Exact Test will be applied for values below five in four-sided tables. The conformity of quantitative data to normal distribution will be tested with Kolmogorov-Simirnov and Shapiro Wilk tests. For statistical analysis of quantitative data in independent groups, Unpaired t test and One-Way Anova test (post hoc Tukey test) will be used for data conforming to normal distribution, Mann-Whitney U, Kruskall-Wallis test will be used for data not conforming to normal distribution and Pearson Correlation coefficient will be used to show the relationship between variables. Statistical significance of the difference was accepted as p<0.05.

Date:11.04.2024 Version No: 01